CLINICAL TRIAL: NCT01056900
Title: An Investigator-sponsored Trial for Observation of the Result After Chondron (Autologous Chondrocytes) Treatment
Brief Title: Observation of the Result After Chondron (Autologous Chondrocytes) Treatment
Status: Completed | Type: Observational
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Nam Yong, Choi, St.Paul Hospital of Catholic University
Other Study IDs: 05CON
Record Dates: First submitted 2010-01-21; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Articular Cartilage Defects of Knee
Keywords: articular cartilage defects; ACI; Autologous Chondrocyte Implantation; Knee joint; chondron

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chondron Implantation: This clinical trial was a follow-up study involving 127 patients from 10 hospitals, for whom autologous chondrocyte transplantation was already performed. All the subjects were investigated as a single group
  Interventions: Procedure: Autologous Chondrocyte Implantation

INTERVENTIONS:
Procedure: Autologous Chondrocyte Implantation — * Test drug: Chondron (more than 12 million chondrocytes in 0.4ml, i.e. 1 vial)
  * Directions and dosage:
  Suspend the cells in the vial sufficiently, and implant them in the defective part, making sure that sufficient amounts are injected.
  Other Names: Chondron(671500010 [ A74600011 ])

SUMMARY:
This investigator-sponsored trial attempts to evaluate the effectiveness of Chondron transplantation by tracking subjects who had the Chondron implantation to observe effectiveness.

DETAILED DESCRIPTION:
Many treatment cases proved that autologous chondrocyte transplantation is a useful treatment method for patients with damaged articular cartilage.

This investigator-sponsored trial attempts to evaluate the effectiveness of Chondron(autologous chondrocyte) transplantation by tracking subjects who had the Chondron implantation to observe effectiveness.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adult males and females aged between 15 and 65
  2. Patients with a partial cartilaginous defect in the ankle joint confirmed arthroscopically or visually
  3. Patients with misalignment between tibia and talus of the ankle joint, lateral ankle instability, and a bony defect in the cartilaginous defect or who had a correction simultaneously or in advance
  4. Patients whose surrounding cartilage is normal
  5. Subjects who consented to the clinical trial or on whose behalf a person with parental rights consented to the clinical trial
* Exclusion Criteria:

  1. Patients hypersensitive to bovine protein
  2. Patients hypersensitive to antibiotics like gentamicin
  3. Patients with inflammatory arthritis, such as rheumatoid arthritis and gouty arthritis
  4. Patients with arthritis associated with autoimmune diseases
  5. Patients who are pregnant, nursing a baby or likely to get pregnant
  6. Patients with other diseases including tumors except for cartilaginous defects of joints
  7. Patients with an anamnesis within the past two years, such as radiation treatment and chemotherapy
  8. Diabetics (however, patients who were normal in the blood glucose test and have no complication due to diabetes will be excluded if the doctor says Chondron can be administered to them)
  9. Patients with infections who are taking antibiotics and antimicrobial agents
  10. Patients who are treated with adrenal cortical hormones
  11. Patients whom the investigators find to be unfit for this clinical trial, such as mental patients

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this exploratory clinical trial Chondron (autologous chondrocytes) is transplanted in the cartilaginous defects and the effectiveness is observed through follow-up. Target subjects are about 5% of about 2,000 patients with Chondron implants.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change of KSS(Knee Society Score)-A,B | pre-operation, post -operation 4month, post-operation 12month, over post-operation 24month.

SECONDARY OUTCOMES:
Additional treatment related to autologous chondrocyte implantation | post -operation 4month, post-operation 12month, over post-operation 24month.
Satisfaction of patients | post -operation 4month, post-operation 12month, over post-operation 24month.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Yong Choi, Principal Investigator — St. Paul Hospital of Catholic Medical College
Locations (1):
- Sewon Cellontech, Sungdong-ku, Seoul, South Korea